CLINICAL TRIAL: NCT04776525
Title: Sequential Neoadjuvant Ifosfamide and Doxorubicin in Localized High-grade Soft Tissue Sarcoma of Extremities and Trunk Wall
Brief Title: Sequential Neoadjuvant Chemotherapy in Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Kjetil Boye, Senior Consultant, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 44-2020
Record Dates: First submitted 2021-02-19; First posted 2021-03-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Soft Tissue Sarcoma
Keywords: Doxorubicin; Ifosfamide; Sarcoma; Neoadjuvant; Sequential
MeSH Terms: conditions — Sarcoma | interventions — Ifosfamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sequential ifosfamide and doxorubicin (Experimental): Four cycles ifosfamide 9 g/m2 and four cycles doxorubicin 80 mg/m2. Each cycle has a duration of 14 days.
  Interventions: Drug: Ifosfamide; Drug: Doxorubicin

INTERVENTIONS:
Drug: Ifosfamide — 3 g/m2 each day for three days
  Other Names: Holoxan
Drug: Doxorubicin — 80 mg/m2 over four hours day 1
  Other Names: Adriamycin

SUMMARY:
Nearly half of patients with high-grade, localized soft tissue sarcoma (STS) of extremities and trunk wall develop disease recurrence after local therapy. Adjuvant chemotherapy with ifosfamide and doxorubicin may improve long-term disease-free survival, but the benefit of adjuvant treatment is limited and predictive factors for treatment response are lacking. The aim of this study is to explore sequential treatment with ifosfamide and doxorubicin in a neoadjuvant setting and to investigate biomarkers predictive of treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of informed consent.
2. Histological diagnosis of soft tissue sarcoma belonging to one of the following histotypes:

   1. Leiomyosarcoma
   2. Malignant peripheral nerve sheath tumor
   3. Undifferentiated pleomorphic sarcoma
   4. Myxofibrosarcoma
   5. Synovial sarcoma
   6. Pleomorphic liposarcoma
   7. Pleomorphic rhabdomyosarcoma
   8. Unclassified spindle cell sarcoma
3. Malignancy grade ≥ 2 according to the Fédération Nationale des Centres de Lutte Contre le Cancer (FNCLCC) grading system.
4. Tumor localized in extremity, girdle and/or trunk wall.
5. Primary tumor size ≥5.0 cm as measured in the longest diameter on diagnostic MRI or CT scan.
6. Primary tumor location below the superficial fascia or involving the superficial fascia, i.e. deep-seated according to the World Health Organization (WHO) Classification of Tumors of Soft Tissue and Bone (4th edition, 2013).
7. The primary tumor must be available for biopsy collection at protocol inclusion.
8. Patients must have a measurable tumor according to RECIST v1.1.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
10. Before patient registration, written informed consent must be given according to national and local regulations.
11. Adequate organ function and bone marrow reserve as indicated by the following laboratory assessments:

    1. Hemoglobin ≥ 8.0 g/dL
    2. Neutrophil count ≥ 1.0 x 109/L
    3. Platelet count ≥ 75 x 109/L
    4. Total bilirubin ≤ 1.5 x the upper limit of normal (ULN)
    5. Creatinine clearance ≥ 60 ml/min based on Cockcroft Gault estimation or direct measurement
12. Negative Hepatitis B and C and HIV serology.
13. Adequate contraception in women of childbearing potential (WOCBP) and their fertile partners during the study and until 6 months after end of study treatment. WOCBP should have a negative highly sensitive serum or urine pregnancy test within 72 hours prior to receiving the first dose of study medication. A woman is considered fertile following menarche and until becoming post-menopausal unless permanently sterile. WOCBP should be willing to use one of the mentioned highly effective methods of birth control mentioned below or be surgically sterile, or abstain from heterosexual activity for the course of the study through 1 year after the last dose of study medication. Methods considered as highly effective birth control methods include combined (estrogen and progestogen containing) or progestogen-only hormonal contraception associated with inhibition of ovulation (oral, intravaginal, injectable, implantable or transdermal), intrauterine device (including hormone-releasing), male condom, bilateral tubal occlusion, vasectomised partner or sexual abstinence (see appendix 5 for definitions).

Exclusion Criteria:

1. Any prior therapy for soft tissue sarcoma.
2. Locoregional or distant metastasis as assessed by CT and/or MRI at time of diagnosis. Patients with lung nodules <10 mm of uncertain etiology may be included.
3. Clinical evidence of serious coagulopathy. Prior arterial/venous thrombosis or embolism does not exclude patients from inclusion, unless patient is considered unfit by study oncologist.
4. Urinary obstruction.
5. Known hypersensitivity towards ifosfamide, doxorubicin or pegfilgrastim, their metabolites and other ingredients in the drug administration formulation.
6. New York Heart Association class II-IV heart disease, myocardial infarction within 6 months of diagnosis of soft tissue sarcoma, active ischemia or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia requiring therapy, uncontrolled hypertension or congestive heart failure.
7. Left ventricular ejection fraction (LVEF) < 50%.
8. Patients with a prior or concurrent malignant disease whose natural history or treatment have the potential to interfere with the safety or efficacy assessment of this clinical trial are not eligible. Patients with a history of breast cancer, requiring continued hormonal treatment (e.g. anti-estrogen or an aromatase inhibitor) may be included. Patients with a history of prostate cancer, requiring continued support with luteinizing hormone releasing hormone (LHRH) agonists, with or without androgens, may be included.
9. Patients not able to give an informed consent or comply with study regulations as deemed by study investigator.
10. Any other significant comorbidities, such as active infection, uncontrolled pulmonary or liver disease, active cystitis, or any other condition, that based on the assessment of the treating physician could compromise compliance with the protocol or predispose the patient to safety risks.
11. Pregnant or lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2036-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 16 weeks
  Partial or complete response using RECIST v1.1

SECONDARY OUTCOMES:
Incidence of treatment-related adverse events as assessed by CTCAE v5.0 and dose reductions (safety and tolerability) | Until 30 days after last dose of study treatment
  Number and type of adverse events, serious adverse events, dose reductions and discontinuation due to toxicity
Correlation between TP53 mutation assessed by sequencing of tumor DNA and overall response | Up to 16 weeks
  To investigate if TP53 mutations assessed by sequencing of tumor DNA predict response to high-dose alkylating chemotherapy and/or sequential doxorubicin monotherapy in STS

OTHER OUTCOMES:
Disease-free survival | Up to 10 years after completion of study treatment
Overall survival | Up to 10 years after completion of study treatment
Health-related quality of life | Up to 10 years after completion of study treatment
  To assess change from baseline in the European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) scores during treatment
Number of patients who experience a change in the extent of the planned surgical procedure due to study treatment | From baseline and up to 6 months
  To investigate if the extent of the surgical procedure is changed due to neoadjuvant treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kjetil Boye, MD PhD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No